CLINICAL TRIAL: NCT05939492
Title: Determining the Feasibility, Acceptability, and Effectiveness of a Self-Guided Mindfulness-Based Intervention in Pediatric Patients With Idiopathic Chest Pain: A Pilot Study
Brief Title: Mindfulness for Pediatric Chest Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Shubhayan Sanatani, Head Division of Cardiology; Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H23-00137
Record Dates: First submitted 2023-06-22; First posted 2023-07-11 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Chest Pain
Keywords: Pediatrics; Idiopathic; Chest Pain
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Intervention Model Description: After a 2-week wash-in period, study participants will be randomly assigned to either the standard of care control group or the mindfulness-based intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Control (No Intervention): Participants in this arm will receive the standard of care. For patients with idiopathic chest pain, the standard of care is typically just reassurance of the benign nature of their pain.
- Mindfulness-Based Intervention (Experimental): Participants in this arm will partake in a 30 day mindfulness-based intervention on the mobile app Headspace.
  Interventions: Behavioral: Mindfulness-Based Intervention

INTERVENTIONS:
Behavioral: Mindfulness-Based Intervention — Participants in the mindfulness-based intervention (MBI) group will be asked to use the Headspace app to sequentially complete the "Basics", "Basics 2", and "Basics 3" courses. Each of these courses lasts 10 days, and participants have the ability to choose how long daily sessions last. Participants can choose between 3, 5, or 10-minute sessions for the "Basics" course; 10 or 15-minute sessions for the "Basics 2" course; and 10, 15, or 20-minute sessions for the "Basics 3" course. These daily sessions are audio recordings that prompt users to engage in a variety of mindfulness techniques, including focusing on their body and breathing, as well as acknowledging thoughts and emotions in a non-judgmental manner.
  Arms: Mindfulness-Based Intervention

SUMMARY:
The goal of this clinical trial is to test mindfulness practices in children with idiopathic chest pain, which is chest pain that does not have a known cause. The main question this study aims to answer is whether children who experience idiopathic chest pain are able to follow a mindfulness program. This study also aims to determine whether mindfulness affects the way children with idiopathic chest pain cope, and if it affects their stress levels, quality of life, frequency of chest pain episodes, and chest pain intensity.

Participants will:

* Complete a survey at the beginning of the study that asks questions about their sex, ethnicity, and history of chest pain and other chronic pains.
* Complete a short survey every day for the entirety of the study that asks about the number, intensity, and duration of chest pain episodes experienced that day.
* Complete 4 surveys, 2 weeks after they have been enrolled in the study: pain coping survey, perceived stress survey, quality of life survey, and mindfulness survey.
* Be randomly placed into either the control group or the mindfulness-based intervention group, 2 weeks after they have been enrolled in the study.
* Receive the standard of care for children with idiopathic chest pain, if they are placed into the control group.
* Use the mobile app Headspace to complete daily mindfulness sessions for the remaining 30 days of the study (starting after the initial 2 week period), if they are placed in the mindfulness-based intervention group.
* Complete 4 surveys at the end of the study: pain coping survey, perceived stress survey, quality of life survey, and mindfulness survey.
* Complete a mindfulness program evaluation survey at the end of the study, only if they are in the mindfulness-based intervention group.

Researchers will collect information from Headspace to see how well participants in the mindfulness-based intervention group are able to follow the mindfulness program. This will help guide future, larger studies that look at the effects of mindfulness-based interventions in children with idiopathic chest pain. Researchers will also compare survey results between the control group and the mindfulness-based intervention group to see if the mindfulness program affects the way children with idiopathic chest pain cope, as well as their stress levels, quality of life, frequency of chest pain episodes, and chest pain intensity.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose primary complaint is recurrent chest pain that is diagnosed as idiopathic or musculoskeletal by a pediatric cardiologist.
* No acute illness.
* Normal ECG.
* Willing and able to download and use the Headspace application on a daily basis.
* Able to complete surveys in the English language.

Exclusion Criteria:

* Patients whose chest pain is secondary to pericarditis, arrhythmia, or structural heart disease.
* Patients with concurrent symptoms that could potentially interfere with the ability to determine the effect on their chest pain (e.g., palpitations or dizziness).
* Unable to provide informed assent.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Participant Recruitment Rate | Baseline (0 days)
  The number of patients who consent to participate in the study compared to the number of patients approached about study participation.
Feasibility: Participant Retention Rate | 44 days
  The number of participants who remain enrolled in the study for the entirety of the study duration compared to the number of participants who consent to participate in the study.
Feasibility: Mindfulness-Based Intervention Program Adherence | 44 days
  Data regarding mindfulness-based intervention program adherence will be collected from Headspace. This includes information about all sessions and length of sessions.
Acceptability: Mindfulness-Based Intervention Program Evaluation | 44 days
  Data regarding mindfulness-based intervention program evaluation will be collected from the mindfulness program evaluation survey. This survey inquires about duration of the mindfulness program and of daily sessions. It also asks about what participants find most and least useful in the program, as well as what participants want more or less of.
Feasibility: Survey Response Rate | 44 days
  The number of surveys completed by participants compared to the number of surveys sent out to be completed.

SECONDARY OUTCOMES:
Pain Coping Strategies | 14 days and 44 days
  Pain coping strategies will be assessed by having participants complete the Pediatric Quality of Life Inventory Pediatric Pain Coping Inventory (PedsQL PPCI).
  This questionnaire is comprised of 41 items, with scores transformed on a scale from 0 (never) to 2 (often). The minimum score is 0 and the maximum is 82. A higher score indicates a greater use of pain coping strategies.
Perceived Stress | 14 days and 44 days
  Perceived stress will be assessed by having participants complete the Perceived Stress Scale (PSS-10).
  This questionnaire is comprised of 10 items. The minimum score is 0 and the maximum is 40. A higher score indicates a higher level of perceived stress.
Patient Quality of Life | 14 days and 44 days
  Quality of life will be assessed by having participants complete the Pediatric Quality of Life Inventory (PedsQL) Generic Core Scale.
  This questionnaire is comprised of 23 items which are reverse scored and linearly transformed to a 0-100 scale as follows:
  0 (never) = 100
  1. (almost never) = 75
  2. (sometimes) = 50
  3. (often) = 25
  4. (almost always) = 0
  The minimum score is 0 and the maximum is 2300. A higher score indicates a better health-related quality of life.
Chest Pain Episode Frequency | Begin at 0 days, daily up to 44 days
  Frequency of chest pain episodes will be assessed by having participants complete the chest pain episodes survey that inquires about how many chest pain episodes they had that day.
Chest Pain Episode Intensity | Begin at 0 days, daily up to 44 days
  Intensity of chest pain episodes will be assessed by having participants complete the chest pain episodes survey that inquires about the average intensity of chest pain episodes they had that day. Intensity will be rated using the Wong-Baker FACES Pain Rating Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Shubhayan Sanatani, MD, Principal Investigator — British Columbia Children's Hospital
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada